CLINICAL TRIAL: NCT06680128
Title: A 2-Stage, Phase I/II, Active-controlled, Randomized, Observer-blinded, Dose-finding Study to Assess the Safety, Reactogenicity, and Immunogenicity of SK Japanese Encephalitis mRNA Vaccines (GBP560) in Healthy Adults (Aged 18 Years and Older)
Brief Title: A Study to Assess the Safety, Reactogenicity, and Immunogenicity of SK Japanese Encephalitis Messenger Ribonucleic Acid (mRNA) Vaccines (GBP560) in Healthy Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GBP560_001
Record Dates: First submitted 2024-10-28; First posted 2024-11-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Japanese Encephalitis Virus Disease
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Stage 1: sequential, Stage 2 : parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Test group 1-1 (GBP560-A) (Experimental): Low dose level(3µg) for GBP560-A in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-A
- Test group 1-2 (GBP560-B) (Experimental): Low dose level (3µg) for GBP560-B in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-B
- Test group1-3 (GBP560-A) (Experimental): Mid dose level (15µg) for GBP560-A in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-A
- Test group1-4 (GBP560-B) (Experimental): Mid dose level (15µg) for GBP560-B in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-B
- Test group1-5 (GBP560-A) (Experimental): High dose level (50µg) for GBP560-A in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-A
- Test group1-6 (GBP560-B) (Experimental): High dose level (50µg) for GBP560-B in stage 1. Participants will receive 2 doses of one of the test vaccines at 4-week intervals, respectively.
  Interventions: Biological: GBP560-B
- Control group1 (IXIARO®) (Active Comparator): Participants will receive 2 doses of one of the active comparators (IXIARO®, 6 Antigen Unit, corresponding to a potency of ≤ 460 ng ED) at 4-week intervals, respectively in Stage 1 and Stage 2.
  Interventions: Biological: IXIARO
- Control group2 (IMOJEV®) (Active Comparator): Participants will receive 1 dose of placebo saline and 1 dose of another active comparator (IMOJEV®, 4.0 - 5.8 log PFU) at 4-week intervals, respectively in Stage 1 and Stage 2.
  Interventions: Biological: IMOJEV; Biological: Normal Saline (Placebo)
- Test group 2-1 (GBP560-A or B) (Experimental): Participants will receive 2 intramuscular injections of the test vaccines in stage 2.
  1st will be on Visit 2 and 2nd will be on Visit 5, in line with the selected dose regimen in stage 1.
  Interventions: Biological: GBP560-A; Biological: GBP560-B
- Test group 2-2 (GBP560-A or B) (Experimental): Participants will receive 2 intramuscular injections of the test vaccines in stage 2.
  1st will be on Visit 2 and 2nd will be on Visit 5, in line with the selected dose regimen in stage 1.
  Interventions: Biological: GBP560-A; Biological: GBP560-B

INTERVENTIONS:
Biological: GBP560-A — injection volume of 0.5mililiter (mL) with each dose on V2(1day) and V5 (29day) in stage1 and stage2.
  Low dose: 3μg Mid dose: 15μg High dose: 50μg
  Arms: Test group 1-1 (GBP560-A); Test group 2-1 (GBP560-A or B); Test group 2-2 (GBP560-A or B); Test group1-3 (GBP560-A); Test group1-5 (GBP560-A)
Biological: GBP560-B — injection volume of 0.5mL with each dose on V2(1day) and V5 (29day) in stage1 and stage2.
  Low dose: 3μg Mid dose: 15μg High dose: 50μg
  Arms: Test group 1-2 (GBP560-B); Test group 2-1 (GBP560-A or B); Test group 2-2 (GBP560-A or B); Test group1-4 (GBP560-B); Test group1-6 (GBP560-B)
Biological: IXIARO — injection volume of 0.5mL on V2(1day) and V5 (29day) in stage1 and stage2
  Arms: Control group1 (IXIARO®)
Biological: IMOJEV — injection volume of 0.5mL on V5 (29day) in stage1 and stage2
  Arms: Control group2 (IMOJEV®)
Biological: Normal Saline (Placebo) — injection volume of 0.5mL on V2 (1day) in stage1 and stage2 (This is for IMOJEV placebo)
  Arms: Control group2 (IMOJEV®)

SUMMARY:
This is a 2-Stage, Phase I/II Study to Assess the Safety, Reactogenicity, and Immunogenicity of SK Japanese Encephalitis mRNA Vaccines (GBP560) in Healthy Adults (Aged 18 Years and Older)

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of SK Japanese Encephalitis mRNA vaccines (GBP560) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

[Age]

1. For Stage 1, participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.

   For Stage 2, participant must be 18 years of age and older, at the time of signing the informed consent.

   [Type of Participant and Disease Characteristics]
2. Participants who are healthy as determined by medical evaluation including medical history, vital signs, physical examination, clinical laboratory tests and medical judgement of the investigator.
3. Participants who are willing and able to attend all scheduled visits and comply with all study procedures.
4. Body mass index (BMI) within the range of 18.5-29.9 kg/m2 (inclusive) at screening

   [Sex and Contraceptive/Barrier Requirements]
5. All participants must agree to be heterosexually inactive or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the 1st study vaccination to 12 weeks after the last study vaccination (Visit 9) (See Appendix 10.4 for detailed contraceptive methods).
6. Female participants with a negative urine or serum pregnancy test at screening.

   * Female participants who are surgically sterile (e.g., having undergone a full hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal with amenorrhea for at least 12 months are not subject to a pregnancy test.

   [Informed Consent]
7. Participants who are capable of giving signed informed consent as described in Appendix 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol before initiation of any trial-specific procedures.

Exclusion Criteria:

[Medical Conditions]

1. Any clinically significant respiratory symptoms (e.g., cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 24 hours prior to the 1st study vaccination. Prospective participants with these conditions cannot be included until 24 hours after resolution.
2. History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease.
3. Any positive test results for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening.
4. History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination in the investigator's opinion.
5. History of hypersensitivity and severe allergic reaction (e.g., anaphylaxis, Guillain-Barre syndrome) to any vaccines or components of the study intervention.
6. History of myocarditis, pericarditis or myopericarditis (including the screening 12-lead ECG results from Stage 1 participants), as assessed by the investigator, indicating probable or possible myocarditis, pericarditis, or myopericarditis, or demonstrating clinically significant abnormalities that could affect participant safety or the interpretation of study findings.
7. History of JEV infection/other flaviviruses infection (e.g., Dengue, West Nile, Zika, St. Louis Encephalitis, Yellow fever).
8. History of malignancy within 1 year prior to the 1st study vaccination (with the exception of malignancy with minimal risk of recurrence at the discretion of the investigator).
9. Significant unstable chronic or acute illness that, in the opinion of the investigator, might pose a health risk to the participant if enrolled, or could interfere with the protocol-specified activities, or interpretation of study results.

   * The AESIs as outlined in Section 8.1.4 should be considered for evaluating the participant
10. Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions).
11. Female participants who are pregnant or breastfeeding.
12. (Only for Stage 1) Current smoker or a recent smoking history within 12 weeks prior to screening. Occasional smoker who smokes up to 10 cigarettes per month may be allowed to participate at the investigator's discretion.

    [Prior/Concomitant medication]
13. Receipt of JEV vaccination/other flaviviruses vaccination in the past.
14. Receipt of any vaccine within 4 weeks prior to the 1st study vaccination or planned receipt of any vaccine from enrollment through 4 weeks after the last study vaccination (Visit 8), except for inactivated influenza vaccination, which may be received at least 2 weeks prior to the 1st study vaccination.
15. Receipt of immunoglobulins and/or any blood or blood-derived products within 12 weeks prior to the 1st study vaccination.
16. Receipt of immunosuppressive therapy, such as any use of anti-cancer chemotherapy or radiation therapy; or systemic corticosteroid therapy (≥10 mg prednisone/day or equivalent) within 12 weeks prior to the 1st study vaccination. The use of inhaled, topical, or nasal glucocorticoid will be permitted.

    [Prior/Concurrent Clinical Study Experience]
17. Participation in another clinical study and receipt of study intervention within 4 weeks prior to the 1st study vaccination, or concurrent, planned participation in another clinical study with study intervention during this study period.

    [Other Exclusions]
18. Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
19. Donation of ≥ 450mL (milliliter) of blood product within 4 weeks prior to screening, or planned donation of blood product from enrollment through 12 weeks after the last study vaccination (Visit 9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing any immediate reactions | 30 minutes (2 hours for the sentinel participants in stage 1) post each vaccination
  For all cohort
Percentage of participants reporting any solicited local Adverse Event (AE) | during the 7 days following each study vaccination
  For all cohort
Percentage of participants reporting any solicited systemic Adverse Event (AE) | during the 7 days following each study vaccination
  For all cohort
Percentage of participants experiencing any unsolicited Adverse Event (AE) | during the 28 days following each study vaccination
  For all cohort
Percentage of participants with any Medically Attended Adverse Event (MAAE) | until 6 months following the last study vaccination
  For all cohort
Percentage of participants experiencing any Adverse Event of Special Interest (AESI)s, AEs leading to study withdrawal and Serious Adverse Event (SAE)s during the entire study period | up to 12 months for stage 1 and up to 24 months for stage 2
  For all cohort
Seroprotection rate for both the respective and cross Japanese encephalitis virus (JEV) strains of each vaccine (SA14-14-2 and Beijing-1 strain) in live-virus neutralizing antibody titers at each time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, 12 months, and 24 months following the 2nd study vaccination.
  For stage 2
Seroresponse rate for both the respective and cross JEV strains of each vaccine (SA14-14-2 and Beijing-1 strain) in live-virus neutralizing antibody titers, from baseline to each subsequent time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, 12 months, and 24 months following the 2nd study vaccination
  For Stage 2
Geometric Mean Titer (GMT) of neutralizing antibody against both the respective and cross JEV strains of each vaccine (SA14-14-2 and Beijing-1 strain) measured by a live-virus neutralization assay (PRNT) at each time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, 12 months, and 24 months following the 2nd study vaccination.
  For stage 2
Geometric mean fold rise of neutralizing antibody against both the respective and cross JEV strains of each vaccine (SA14-14-2,Beijing-1 strain), measured by a live-virus neutralization assay(PRNT), from each pre-vaccination to each subsequent timepoint | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, 12 months, and 24 months following the 2nd study vaccination
  For Stage 2
Geometric mean fold reduction of neutralizing antibody against both respective and cross JEV strains of each vaccine (SA-14-14-2,Beijing-1 strain), measured by live-virus neutralization assay (PRNT) from persistence baseline to each subsequent timepoint | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, 12 months, and 24 months following the 2nd study vaccination.
  For Stage 2

SECONDARY OUTCOMES:
Seroprotection rate for both the respective and cross JEV strains of each vaccine (SA14-14-2 and Beijing-1 strain) in live-virus neutralizing antibody titers at each time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination
  For Stage 1
Seroresponse rate for both the respective and cross JEV strains of each vaccine (SA14-14-2 and Beijing-1 strain) in live-virus neutralizing antibody titers, from baseline to each subsequent time point. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination
  For stage 1
GMT of neutralizing antibody against both the respective and cross JEV strains of each vaccine (SA14-14-2 and Beijing-1 strain) measured by a live-virus neutralization assay (PRNT) at each time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination
  For stage 1
Geometric mean fold rise of neutralizing antibody against both the respective and cross JEV strains of each vaccine (SA14-14-2,Beijing-1 strain), measured by live-virus neutralization assay(PRNT), from each pre-vaccination to each subsequent timepoint | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For stage 1
Geometric mean fold reduction of neutralizing antibody against both respective and cross JEV strains of each vaccine (SA-14-14-2,Beijing-1 strain),measured by live-virus neutralization assay(PRNT) from persistence baseline to each subsequent timepoint | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination.
  For Stage1
Cell-mediated response for cytokines expressed by Cluster of Differentiation 4+ Cluster of Differentiation 8+ T cells (Interferon-γ, Tumor Necrosis Factor-α, measured by Fluorescence-Activated Cell Sorting-Intracellular Cytokine Staining assay. | At baseline, 4 weeks following the 1st study vaccination, and at 4 weeks and 6 months following the 2nd study vaccination
  For all cohort

OTHER OUTCOMES:
Seroprotection rate for the heterologous JEV strains of each vaccine (including, but not limited to K95A07, Bennett, JKT 6468, Sangju-v1 strains) in live-virus neutralizing antibody titers at each timepoint. | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination. and 24 months following the 2nd study vaccination (for stage2 only)
  will be evaluated exclusively in a subset of approximately 20% of participants in stage 1, 10% of participants in stage 2
GMT of neutralizing antibody against the heterologous JEV strains of each vaccine (including, but not limited to K95A07, Bennett, JKT 6468, Sangju-v1 strains) measured by a live-virus neutralization assay (PRNT) at each timepoint | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination. and 24 months following the 2nd study vaccination (for stage2 only)
  will be evaluated exclusively in a subset of approximately 20% of participants in stage 1, 10% of participants in stage 2
Seroresponse rate for the heterologous JEV strains of each vaccine (including, but not limited to K95A07, Bennett, JKT 6468, Sangju-v1 strains) in live-virus neutralizing antibody titers, from baseline to each subsequent time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination. and 24 months following the 2nd study vaccination (for stage2 only)
  will be evaluated exclusively in a subset of approximately 20% of participants in stage 1, 10% of participants in stage 2
Geometric mean fold rise of neutralizing antibody against the heterologous JEV strains of each vaccine (including,but not limited to K95A07, Bennett, JKT 6468, Sangju-v1) measured by the PRNT assay, from each pre-vaccination to each subsequent time point | At baseline, 2 weeks, 4 weeks following the 1st study vaccination, and at 2 weeks, 4 weeks, 3 months, 6 months, and 12 months following the 2nd study vaccination. and 24 months following the 2nd study vaccination (for stage2 only)
  will be evaluated exclusively in a subset of approximately 20% of participants in stage 1, 10% of participants in stage 2.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Nucleus Network - Brisbane (Q Pharm), Brisbane
  - Nucleus Network - Melbourne, Melbourne
- New Zealand Clinical Research, Christchurch, Central City, New Zealand

IPD SHARING:
Plan to Share IPD: No